CLINICAL TRIAL: NCT01520207
Title: Pilot Study of Intravenous Mannitol During Hemodialysis Initiation to Reduce the Occurrence of Intra-dialytic Hypotension.
Brief Title: Mannitol - Potential Role in Hemodialysis Initiation for Reduction of Intra-dialytic Hypotension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Sushrut S Waikar, Associate Professor of Medicine, Harvard Medical School, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: NCT01520207
Record Dates: First submitted 2012-01-25; First posted 2012-01-27 (Estimated); Results first posted 2017-10-19 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Intra-dialytic Hypotension
MeSH Terms: interventions — Mannitol; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo group: (0.9% normal saline) (Placebo Comparator): 0.9% saline will be administered (IV) during the hemodialysis session at 1.25mL/kg/hour (max 375mLs per session). Administration will be discontinued 30 minutes before the end of the hemodialysis session.
  Interventions: Drug: 0.9% saline
- Intervention: intravenous mannitol (20%) (Active Comparator): Mannitol will be administered (IV) during the hemodialysis session at a maximum rate of 0.25g/kg/hour (maximum rate 25g/hour; maximum 75g per session; maximum volume 375mLs per session). Administration will be discontinued 30 minutes before the end of the hemodialysis session.
  Interventions: Drug: Mannitol (20%)

INTERVENTIONS:
Drug: Mannitol (20%) — 0.25g/kg/hour (maximum rate 25g/hour; maximum 75g per session; maximum volume 375mLs per session)
  Arms: Intervention: intravenous mannitol (20%)
Drug: 0.9% saline — 1.25mL/kg/hour; maximum 125mLs/hour; maximum total volume 375mLs per treatment
  Arms: Placebo group: (0.9% normal saline)

SUMMARY:
Kidney failure can result from a variety of conditions and can be temporary or permanent. Hemodialysis is available as a replacement treatment to perform the work that the kidneys normally do. However, the dialysis procedure can be associated with rapid changes in the composition of the blood - this may lead to changes in blood pressure and in turn reduced blood supply to important parts of the body. We aim to investigate if giving a medicine (called mannitol) during dialysis may be able to reduce the frequency of these low blood pressure events.

ELIGIBILITY:
Inclusion Criteria:

* Renal failure requiring intermittent hemodialysis initiation; adult patients aged over 18 years; written informed consent

Exclusion Criteria:

* Hyponatremia <130 mmol/L; acute myocardial infarction or stroke in previous 7 days; cardiac transplant; ventricular arrhythmia; unstable angina; use of pressors/midodrine; enrollment in conflicting research study; institutionalized individuals; pregnancy; prisoners; documented allergy to mannitol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sushrut S Waikar, MD, MPH, Principal Investigator — Brigham and Women's Hospital, Harvard Medical School; Finnian R Mc Causland, MB, MMSc, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Curtis KA, Waikar SS, Mc Causland FR. Higher NT-proBNP levels and the risk of intradialytic hypotension at hemodialysis initiation. Hemodial Int. 2024 Jan;28(1):77-84. doi: 10.1111/hdi.13125. Epub 2023 Oct 24. PMID 37875429
- [Derived] Mc Causland FR, Claggett B, Sabbisetti VS, Jarolim P, Waikar SS. Hypertonic Mannitol for the Prevention of Intradialytic Hypotension: A Randomized Controlled Trial. Am J Kidney Dis. 2019 Oct;74(4):483-490. doi: 10.1053/j.ajkd.2019.03.415. Epub 2019 Apr 27. PMID 31040088

RESULTS

PARTICIPANT FLOW:
Recruitment Details: July 2012 - Jul 2016
Period: Overall Study
Arm/Group | Placebo Group: (0.9% Normal Saline) | Intervention: Intravenous Mannitol (20%)
Started | 27 | 25
Completed | 25 | 25
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Group: (0.9% Normal Saline) | Intervention: Intravenous Mannitol (20%) | Total
Number analyzed (Participants) | 27 | 25 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (14.7) | 53.4 (17.4) | 55.6 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 14 | 12 | 26
Region of Enrollment [Number; unit: participants]
  United States | 27 | 25 | 52

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Mannitol Administration in Reducing the Frequency of Intra-dialytic Hypotension (Decline in Systolic Blood Pressure) During the First Three Hemodialysis Initiation Sessions.
Description: SBP decline during first three sessions
Time Frame: First three hemodialysis sessions (5 days)
Population: SBP decline
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo Group: (0.9% Normal Saline) | Intervention: Intravenous Mannitol (20%)
Number analyzed (Participants) | 27 | 25
mmHg | 19 (16) | 15 (11)

ADVERSE EVENTS:
Time Frame: 4 years
Description: Adverse events were monitored for all participants during their HD sessions
Arm/Group | Placebo Group: (0.9% Normal Saline) | Intervention: Intravenous Mannitol (20%)
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/25
Other Adverse Events (participants affected / at risk) | 18/27 | 17/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Group: (0.9% Normal Saline) (N=27) | Intervention: Intravenous Mannitol (20%) (N=25)
Cramps (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2) — Cramps
Hypertension (Cardiac disorders) | 10 (15) | 9 (15) — HTN
Hypotension (Cardiac disorders) | 2 (4) | 2 (2)
Headache (Nervous system disorders) | 2 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (5) | 1 (1)
UTI (Infections and infestations) | 0 (0) | 1 (1)
Access issues (Vascular disorders) | 2 (2) | 2 (2)
Oxygen Requirement (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (7)
Chest Pain (Cardiac disorders) | 0 (0) | 2 (2)
Confusion (Nervous system disorders) | 2 (2) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes